CLINICAL TRIAL: NCT03389490
Title: A Pilot Study to Describe the Glycaemic Variability of Insulin Glargine 300U/ml Versus NPH (Neutral Protamine Hagedorn) in the Insulin-naïve Type 2 Diabetes Patients Following a Patient-adjusted Insulin Algorithm in Hong Kong
Brief Title: Toujeo Versus NPH Self-titration Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elaine Chow (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Elaine Chow, Dr, Clinical Lecturer, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLARGL08588
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin, Isophane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Insulin glargine 300U/ml
  Interventions: Drug: Insulin Glargine 300 UNT/ML
- Control (Active Comparator): Neutral Protamine Hagedorn insulin
  Interventions: Drug: Neutral protamine hagedorn insulin

INTERVENTIONS:
Drug: Insulin Glargine 300 UNT/ML — Self titration of insulin glargine U300
  Arms: Active
Drug: Neutral protamine hagedorn insulin — Self titration of NPH insulin
  Arms: Control

SUMMARY:
This is a 24 week, multicentre, prospective, randomized, controlled, parallel-designed (1:1) pilot study.The study will compare glycemic variability in patients treated with insulin glargine U300/ml insulin versus conventional (NPH) insulin using a self titration algorithm.50 type 2 diabetes patients who are newly started on insulin will be recruited. They will be randomly allocated to either insulin glargine U300 or NPH insulin for 26 weeks. All subjects will follow a insulin-self titration algorithm. The study will consist of 9 visits over 26 weeks. Blood glucose variability will be collected by CGM for 7 consecutive days at baseline (week -1) and at week 24.Secondary endpoints other than data on glycemic variability, including HbA1c, fasting plasma glucose, inflammatory markers will be measured during three periods (week 0, week 12 and week 24).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic suboptimally controlled on their previous antidiabetic treatment

  * 18 ≤ age ≤ 75
  * Stable dose of oral antidiabetic treatment for > 8 weeks
  * The number of OADs that the patients used should be "3" or less
  * HbA1c level > 7.0% and < 10%
  * Fasting plasma glucose > 8mmol/L and <15mmol
  * BMI < 40 kg/m2
  * Patient who is capable and willing to perform regular SMBG
  * Patient who is capable and willing for insulin injection
  * Confirmed written consent
  * Insulin naïve

Exclusion Criteria:

* Participation in a clinical trial with any investigational drug used with curative intent and within 30 days prior to study entry
* Patient known to have hypoglycaemia unawareness or recurrent major hypoglycaemia
* Any product containing prandial insulin
* Concomitant medication known to interface with glucose metabolism (such as systematic steroids)
* Change in dose of non-insulin anti-diabetic treatment or initiation of new anti-diabetic medications in the last 8 weeks prior to screening
* Patients treated with steroid or nonsteroidal anti-inflammatory drugs
* Patient who had experienced an acute concurrent illness during the 3-month period before the investigation
* Patient with hepatic disease and end-stage renal disease
* Patients unable to comply with follow-up visits
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Glycemic variability | 24 weeks
  Standard deviation of glucose from continuous glucose monitoring

SECONDARY OUTCOMES:
Glycemic variability | 24 weeks
  Mean Amplitude of Glycemic excursions and Means of Daily Differences
Percentage time in target | 24 weeks
  Percentage of time <3.0mmol/L and >10.0mmol/L
Glycated haemoglobin | 24 weeks
  HbA1c
Fasting blood glucose | 24 weeks
  FPG
Incidence of hypoglycemia | 24 weeks
  Overall incidence of hypoglycemia and nocturnal hypoglycemia
Proportion of patients achieving HbA1c <7.0% | 24 weeks
  Proportion of patients achieving HbA1c <7.0% at week 24 without confirmed hypoglycemia
Treatment satisfaction | 24 weeks
  ITSQ questionnaire
Inflammatory markers | 24 weeks
  change in hs C reactive protein
Heart rate variability | 24 weeks
  Change in heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ling J, Poon EWM, Yang A, Yeung T, Loo K, Ozaki R, Ma RCW, Luk AOY, Kong APS, Chan JCN, Chow E. Glycemic Variability and Time in Range During Self-titration of Once Daily Insulin Glargine 300 U/ml Versus Neutral Protamine Hagedorn Insulin in Insulin-naive Chinese Type 2 Diabetes Patients. Diabetes Ther. 2021 May;12(5):1399-1413. doi: 10.1007/s13300-021-01046-6. Epub 2021 Mar 18. PMID 33738774
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419